CLINICAL TRIAL: NCT06464107
Title: Endometrial Cancer Cell Collection With the Preprogen PadKit™
Brief Title: Endometrial Cell Collection With the PadKit
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hackensack Meridian Health (Other)
Collaborators: Preprogen (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: Pro2023-0428
Record Dates: First submitted 2024-06-06; First posted 2024-06-18 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Neoplasms
Keywords: endometrial cancer; endometrial hyperplasia; neoplasms; atypical endometrial hyperplasia; Endometrial cells; interlabial pad
MeSH Terms: conditions — Neoplasms; Endometrial Neoplasms; Endometrial Hyperplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Biopsy proven hyperplasia/endometrial cancer with planned hysterectomy (Experimental): Women with biopsy proven hyperplasia/endometrial cancer with planned hysterectomy
  Interventions: Device: PadKit™ from Preprogen
- Benign clinical indications (Experimental): Women with planned hysterectomy for benign clinical indications
  Interventions: Device: PadKit™ from Preprogen

INTERVENTIONS:
Device: PadKit™ from Preprogen — The interlabial pad is classified as a Class 1 device by the FDA and the device is exempt from requiring a 510(k) approval.
  The interlabial pad is worn for 4-6 consecutive hours and collects cells shed from the cervix and uterine cavity. The pad is then removed and placed in the smaller, inner tube that contains the transport solution. After replacing the lid securely, it is then carefully placed back inside the larger outer tube with the outer lid secured and returned to the original box. The entire box is placed in the polybag and mailed back to the lab for analysis.

SUMMARY:
All patients will be provided with a Preprogen Pad to be worn for 4-6 hours to collect cells shed by the endometrium. After the kit is returned to the Preprogen laboratory, a brief survey will be completed. Analysis will be conducted to determine if the PadKit™ can collect a sample of endometrial cells sufficient to differentiate between normal and atypical hyperplasia/malignant cells in blinded samples provided to the laboratory for analysis.

ELIGIBILITY:
Inclusion criteria

1. Women who present to Gynecologic Oncology for surgical intervention and have not undergone prior hysterectomy.

1. Cohort 1: has biopsy proven atypical hyperplasia or endometrial cancer.
2. Cohort 2: women with planned hysterectomy for benign clinical indications

Exclusion criteria

1. Unable to provide informed consent
2. Women who have previously undergone uterine surgery (subtotal, or supracervical hysterectomy).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 80 (Estimated)
Dates: Start 2024-05-31 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Observation of the presence of endometrial cells captured by the pad. | Within 7 days after receipt of the pad from patients
  Direct observation of the absence or presence of endometrial cells on the pad by the pathologist
Association of the presence/absence of cells and morphology | Within 7 days after receipt of the pad from patients
  Analysis for the presence of abnormal histology and morphological classification as normal, hyperplastic, or malignant.

SECONDARY OUTCOMES:
Patient preferences - Comfort | Within the same day and after wearing the pad for 4-6 hours
  To determine patient preferences for using the interlabial PadKit™ vs current standard of care diagnostic tools including transvaginal ultrasound, endometrial biopsy, CT scan, and/or Dilation & Curettage (D&C).
  Patient preferences regarding comfort of wearing the pad are captured using a 1-3 Likert scale with 1 being not comfortable and 3 being comfortable.
Patient preferences - Simplicity of using the pad | Within the same day and after wearing the pad for 4-6 hours
  To determine patient preferences for using the interlabial PadKit™ vs current standard of care diagnostic tools including transvaginal ultrasound, endometrial biopsy, CT scan, and/or Dilation & Curettage (D&C).
  Patient preferences regarding simplicity of using the pad are captured using a 4 Likert scale with 1 being not easy and 4 being very easy.

CONTACTS AND LOCATIONS:
Overall Officials: Mark G Borowsky, MD, Principal Investigator — Hackensack Meridian Health
Locations (2):
- United States (2):
  - Jersey Shore University Medical Center, Neptune City, New Jersey
  - Riverview Medical Center, Red Bank, New Jersey

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] American Cancer Society Endometrial Cancer Statistics. Retrieved from : https://www.cancer.org/cancer/types/endometrial-cancer/about/key-statistics.html
- [Background] Hinson S, Molberg K, Mir M, Flores M, Zheng W, Lucas E. Age cutoff for reporting of benign-appearing endometrial cells in Papanicolaou specimens; should it be raised? A 10-year retrospective study from a large county hospital. J Am Soc Cytopathol. 2019 Mar-Apr;8(2):78-83. doi: 10.1016/j.jasc.2018.09.002. Epub 2018 Sep 11. PMID 31287423
- [Background] Greenspan DL, Cardillo M, Davey DD, Heller DS, Moriarty AT. Endometrial cells in cervical cytology: review of cytological features and clinical assessment. J Low Genit Tract Dis. 2006 Apr;10(2):111-22. doi: 10.1097/01.lgt.0000210130.01016.ad. PMID 16633242
- [Background] Lu KH, Broaddus RR. Endometrial Cancer. N Engl J Med. 2020 Nov 19;383(21):2053-2064. doi: 10.1056/NEJMra1514010. No abstract available. PMID 33207095
- [Background] Pangarkar MA. The Bethesda System for reporting cervical cytology. Cytojournal. 2022 Apr 30;19:28. doi: 10.25259/CMAS_03_07_2021. eCollection 2022. PMID 35673697
- [Background] Sangtani A, Wang C, Weaver A, Hoppman NL, Kerr SE, Abyzov A, Shridhar V, Staub J, Kocher JA, Voss JS, Podratz KC, Wentzensen N, Kisiel JB, Sherman ME, Bakkum-Gamez JN. Combining copy number, methylation markers, and mutations as a panel for endometrial cancer detection via intravaginal tampon collection. Gynecol Oncol. 2020 Feb;156(2):387-392. doi: 10.1016/j.ygyno.2019.11.028. Epub 2019 Nov 28. PMID 31787246